CLINICAL TRIAL: NCT01314820
Title: Effects of Joint Effusion on Quadriceps Muscle in Patients With Knee Osteoarthritis
Brief Title: Effects of Joint Effusion on Quadriceps Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Department of Rehabilitation Medicine, Seoul St. Mary's Hospital,, College of Medicine, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KC09OISI0161
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2010-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Effusion.
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Saline Solution; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal saline injection (Active Comparator): 20 cc normal saline injection into the knee joint
  Interventions: Other: normal saline injection
- sham injection (Sham Comparator): knee injection without saline
  Interventions: Other: sham injection

INTERVENTIONS:
Other: normal saline injection — 20 cc normal saline injection into knee joint
  Other Names: normal saline
  Arms: normal saline injection
Other: sham injection — no saline injection
  Other Names: no normal saline
  Arms: sham injection

SUMMARY:
The present study investigated whether the presence of fluid in the joint affected peak torque and the root mean square (RMS) values of surface electromyography (EMG) in patients symptomatic for osteoarthritis (OA).

DETAILED DESCRIPTION:
Several studies have shown that knee effusion influenced quadriceps muscle activity and induced quadriceps arthrogenic muscle inhibition in normal volunteers. However, the effect of joint effusion on the quadriceps of patients with OA is controversial,and few patients with OA have been included in studies of joint effusion.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or older with knee osteoarthritis
* knee pain without joint effusion confirmed by ultrasonography

Exclusion Criteria:

* the presence of knee joint effusion determined using US
* a history of knee injury or surgery
* a history of knee injection within 3 months
* a history of inflammatory arthritis
* taking anticoagulants
* balance or gait disturbance
* diabetes mellitus

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
the peak torque of the knee extensors | within 5 minutes after intervention
  to evaluate the effect of effusion on the peak torque of the knee extensors

SECONDARY OUTCOMES:
the root mean square values of the vastus medialis and vastus lateralis muscles | within 5 minutes after intervention
  to evaluate the effect of effusion on the RMS of the vastus medialis (VM) and vastus lateralis (VL) muscles

CONTACTS AND LOCATIONS:
Overall Officials: Jongin Lee, M.D, Study Director — Department of Rehabilitation Medicine, Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea
Locations (1):
- Department of Rehabilitation Medicine, Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Fahrer H, Rentsch HU, Gerber NJ, Beyeler C, Hess CW, Grunig B. Knee effusion and reflex inhibition of the quadriceps. A bar to effective retraining. J Bone Joint Surg Br. 1988 Aug;70(4):635-8. doi: 10.1302/0301-620X.70B4.3403614.
- [Background] Jones DW, Jones DA, Newham DJ. Chronic knee effusion and aspiration: the effect on quadriceps inhibition. Br J Rheumatol. 1987 Oct;26(5):370-4. doi: 10.1093/rheumatology/26.5.370. PMID 3664162
- [Background] Rice D, McNair PJ, Dalbeth N. Effects of cryotherapy on arthrogenic muscle inhibition using an experimental model of knee swelling. Arthritis Rheum. 2009 Jan 15;61(1):78-83. doi: 10.1002/art.24168. PMID 19116960